CLINICAL TRIAL: NCT02215421
Title: Kiddio Food Fight: Training Parents in Effective Vegetable Parenting
Brief Title: Mommio: Training in Vegetable Parenting
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding did not allow for completion of game programming
Sponsor: Archimage, Inc. (Industry)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H-33915; R44HD075521 (NIH)
Record Dates: First submitted 2014-08-08; First posted 2014-08-13 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-10

CONDITIONS: Obesity
Keywords: vegetables; dietary intake; preschoolers; parents; video game
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Play Mommio for 2 months (Experimental): The objective is to build parent's skills in encouraging their child to eat vegetables. The player is asked to read a novella, "Totally Frobisher" (providing backstory to the game), and play a game called Mommio (a "casual" video game for parents of 3 to 5 year old children). The player calls Kiddio, the child character, to dinner, and offers a vegetable (V) (selected from among several). Kiddio refuses. The player is offered a selection of V parenting statements (from the scientific literature on food parenting) or manipulation of the environment (e.g. turning off the kitchen TV) to control the situation and encourage the child to eat the V. As problems arise (e.g. a permissive father saying he doesn't like vegetables), the player must select ways to cope. Players set a goal to do with their child at home what they learned in the game. Game episodes include food store shopping, eating in the car, at grandma's, and at a fast food store.
  Interventions: Behavioral: Mommio
- No game play (No Intervention): No intervention control.

INTERVENTIONS:
Behavioral: Mommio — The objective is to build parent's skills in encouraging their child to eat vegetables. The player is asked to read a novella, "Totally Frobisher" (providing backstory to the game), and play a game called Mommio (a "casual" video game for parents of 3 to 5 year old children). The player calls Kiddio, the child character, to dinner, and offers a vegetable (V) (selected from among several). Kiddio refuses. The player is offered a selection of V parenting statements (from the scientific literature on food parenting) or manipulation of the environment (e.g. turning off the kitchen TV) to control the situation and encourage the child to eat the V. As problems arise (e.g. a permissive father saying he doesn't like vegetables), the player must select ways to cope. Players set a goal to do with their child at home what they learned in the game. Game episodes include food store shopping, eating in the car, at grandma's, and at a fast food store.
  Other Names: Kiddio: Food Fight; Kiddia
  Arms: Play Mommio for 2 months

SUMMARY:
A 20 episode video game called Mommio simulates parent-child feeding interactions for parents of 3-5 year old children within a storyline addressing a problem commonly reported by parents (getting their 3-5 yo to taste a vegetable, which is often a first step toward eating the vegetable), thereby training parents in effective food parenting practices. This research evaluates whether the 20 episodes targeting barriers identified by parents across five levels of difficulty influences vegetable parenting practices and children's dietary intake. We had to discontinue the study since changes in commercial availability of game development software required reprogramming and available funding did not allow for completion of game programming. Thus, no game evaluation was possible.

DETAILED DESCRIPTION:
Video games for parents that simulate interactions with a child using a narrative, offering feedback on performance and goal setting for changing practices in the real world, and addressing vegetable (V) feeding problems commonly reported by parents, may elicit desirable cognitive, affective, and behavioral outcomes.

The rationale for training parents of preschool children in effective V parenting practices is that: 1) parents have an important influence on young children's dietary intake; 2) child dietary intake tracks into the adult years; and 3) high V consumption protects against several chronic diseases later in life. Since parents of young children commonly complain about not getting their child to eat V, there should be broad interest in playing Mommio.

A pre-post randomized clinical trial with 110 parents of 3-5 year olds who report having difficulty getting their child to eat vegetables will be employed. The primary outcome will be parent report of children's dietary intake; the secondary outcome will be use of V parenting practices.

We had to discontinue the study since changes in commercial availability of game development software required reprogramming and available funding did not allow for completion of game programming. Thus, no game evaluation was possible.

ELIGIBILITY:
Inclusion Criteria:

* being a parent of a child 3-5 years old
* willing to complete all measures
* having an iPhone.

Exclusion Criteria:

* the parent not speaking English (since the games are in English alone, due to budget constraints);
* having a 3-5 year old child with a medical condition that influences diet; or
* a parent with an illness that impairs the ability to complete questionnaires

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2015-06; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Change in Parent Reported Child Vegetable FFQ | One month from pre to post
  To assess the preschool child's usual vegetable (V) intake, the participating parent will complete the V items from a 36 item FV screener which was demonstrated to have acceptable correlations with serum lycopene, lutein, cryptoxanthin, alphacarotene, and beta-carotene with a validity coefficient (r=0.35 with total carotenoids) comparable to the sum of three 24-hour dietary recalls. Parents have been shown to reliably and validly report preschool child diet intake. The response scales will be worded to reflect child's intake in the previous week. Item responses will be summed to estimate number of V servings consumed in the previous week. This questionnaire has been validated for parent report on children, and was sensitive to change.

SECONDARY OUTCOMES:
Change in Vegetable Parenting Practices Questionnaire | One month from pre to post
  Fruit and Vegetable Parenting Practices Questionnaire (FVPPQ), a parent-report questionnaire, includes 33 items associated with the effectiveness of parenting practices to get children to eat FV. Items will be scored on a three-point scale to indicate frequency of use of V parenting practices (1 - "frequently", 2 - "sometime", 3 - "rarely-never"). Internal consistency has been demonstrated. Helping HAND induced changes in these parenting practices.

OTHER OUTCOMES:
Qualitative Interviews | One month at post only
  The intensive interviews will be conducted using a standardized script and commonly accepted procedures (e.g., 8-10 open ended questions, with follow up questions, prompts, and areas to probe). The questions will assess whether they attempted changes in their vegetable parenting practices with their 3-5 year old child, problems they encountered, what parents liked and disliked about the game, and how it could be made better. The parents' interviews will be about 30 minutes and audio tape recorded. Audio tapes will be transcribed verbatim and checked for accuracy prior to analysis. Following generally accepted qualitative data coding and analysis procedures, NVIVO, a qualitative software analysis program, will be utilized to facilitate data coding, retrieval, and analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Buday, FAIA, Principal Investigator — Archimage, Inc.
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

REFERENCES:
- [Background] Beltran A, O'Connor T, Hughes S, Baranowski J, Nicklas TA, Thompson D, Baranowski T. Alpha Test of a Videogame to Increase Children's Vegetable Consumption. Games Health J. 2012 Jun;1(3):219-222. doi: 10.1089/g4h.2011.0027. PMID 24761315
- [Background] Baranowski T, O'Connor T, Hughes S, Beltran A, Baranowski J, Nicklas T, Sleddens E, Thompson D, Lu AS, Buday R. Smart phone video game simulation of parent-child interactions: Learning skills for effective vegetable parenting. In: Arnab S, Dunwell I, Debattista K (Eds). Serious Games for Healthcare: Applications and Implications. Hershey, PA: IGI Global, 2012, 248-265.